CLINICAL TRIAL: NCT03201172
Title: Prospective Observational 2 Year Follow-up on a Retrospective Cohort of Primary Unicompartmental Knee Arthroplasty (UKA) Patients Treated With Univation® X or iUni®.
Brief Title: Univation® X Follow-Up Study
Status: Completed | Type: Observational
Sponsor: Aesculap AG (Industry)
Responsible Party: Sponsor
Other Study IDs: AAG-O-H-1641
Record Dates: First submitted 2017-05-23; First posted 2017-06-28 (Actual); Last update posted 2021-04-15 (Actual); Status verified 2021-04

CONDITIONS: Unicompartmental Knee Arthroplasty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Univation® X
  Interventions: Device: Primary Unicompartmental Knee Arthroplasty
- iUni®
  Interventions: Device: Primary Unicompartmental Knee Arthroplasty

INTERVENTIONS:
Device: Primary Unicompartmental Knee Arthroplasty — Primary implantation of an unicompartmental knee implant

SUMMARY:
The study is designed as a monocentric, prospective, observational, comparative follow-up study based on two previously treated patient groups. The first group consists of patients treated with the patient-specific unicondylar knee implant iUni®. For that group, 30 patients will be included in the study and analyzed. The final follow-up after 24 months has already been documented by the study center. Compared to that, a consecutive series of 50 Univation® X patients will be invited for a 24 months follow-up in 2018. In total, it is planned to include 80 retrospective patients for that historical control study design.

The products under investigation were used in routine clinical practice and according to the authorized Instructions for Use (IfU). Those data that are obtained in routine clinical use will be documented in the Case Report Form (CRF).

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent UKA in 2015/2016 (using one of the products under investigation)
* Signed informed consent

Exclusion Criteria:

* pregnancy
* patients < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult patients
Sampling Method: Non-Probability Sample
Enrollment: 77 (Actual)
Dates: Start 2017-09-25 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
Knee joint function | 2 years after primary implantation
  Knee Society Score

SECONDARY OUTCOMES:
KOOS | 2 years after primary implantation
  Knee Injury and Osteoarthritis Outcome Score
axis justice position | preoperative and until discharge from hospital (within 1 week postoperatively)
  radiological analysis
radiolucent lines | 2 years after primary implantation
  radiological analysis
tibial slope | 2 years after primary implantation
  radiological analysis

OTHER OUTCOMES:
Adverse Events | 2 years after primary implantation
  Number of Adverse Events during Follow-Up

CONTACTS AND LOCATIONS:
Locations (1):
- St. Vincenz Hospital Brakel, Brakel, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Haaker R, Moussa A, Sabev D. No advantage for patient-specific UKA in comparison with standard UKA regarding clinical and functional results at short-term follow-up. Eur J Orthop Surg Traumatol. 2025 Aug 27;35(1):362. doi: 10.1007/s00590-025-04467-2. PMID 40866508